CLINICAL TRIAL: NCT03144063
Title: Improving the Assessment of Systemic Lupus Erythematosus Disease Activity
Brief Title: Improving the Assessment of SLE Disease Activity
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Zahi Touma, Principal Investigator, University Health Network, Toronto
Other Study IDs: 15-9195
Record Dates: First submitted 2017-04-28; First posted 2017-05-08 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Lupus Erythematosus, Systemic; SLE
Keywords: Disease Activity; SLEDAI-2K
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Toronto Lupus Cohort: Objective 1 and 3 Cohort:
  * ≥4 American College of Rheumatology (ACR) criteria or 3 ACR criteria plus a typical histological lesion of SLE on renal or skin biopsy
  * Clinician's diagnosis based on his/her assessment
  * Patients from the Toronto Lupus Clinic with regular follow-up, defined as having follow up visits at 3 and 6 months from the baseline visit (1st study visit).
- BLISS-52 Cohort: Objective 2 Cohort:
  Validation of the SLEDAI-2KG will be completed on BLISS-52 trial data. The extracted trial data consists of data on all patients that participated in the trial.
- BLISS-76 Cohort: Objective 2 Cohort:
  Validation of the SLEDAI-2KG will be completed on BLISS-76 trial data. The extracted trial data consists of data on all patients that participated in the trial.

SUMMARY:
Physicians' assessment of disease activity in SLE is fundamental but challenging. The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI-2K) is one of the most commonly used disease activity indices. Clinical trials experience suggested that the disease activity instruments did not function well on their own, and composite measures were developed to address this issue. This approach has been adopted after learning from clinical trials that the absence of a robust sensitive index is a major flaw when designing a trial. Another issue with clinical trials is the confounding effect of corticosteroids, which to date have been the most effective treatment for the management of lupus. However, unregulated use of corticosteroids in drug trials decrease the investigator's ability to differentiate between the tested drugs and placebo as they appear to enhance response among the placebo arm and thus mask the effect of the tested drug.

In this study, the aim is to develop and validate a new index, SLEDAI-2K Glucocorticosteroid Index (SLEDAI-2KG). It is very challenging to evaluate improvement in drug trials in the context of the standard of care treatment which includes corticosteroids. This novel index, SLEDAI-2KG, will help to overcome the confounding effect of corticosteroids and to allow for more accurate description of disease improvement and thus facilitate accurate investigations of new therapeutic agents.

DETAILED DESCRIPTION:
Objectives:

1. To describe the development and initial validation of the SLEDAI-2KG using the Toronto Lupus Cohort (TLC) database.
2. To conduct further validation of SLEDAI-2KG using BLISS trial data.
3. To assess concurrent construct validity of SLEDAI-2KG prospectively in the University of Toronto Lupus Clinic.

Study design:

1. Objective one is a single center study aiming to derive a new index, SLEDAI-2KG, based on SLEDAI-2K. Scoring of SLEDAI-2KG will be determined in this study.
2. Objective two is a retrospective analysis conducted on prospectively collected data from two clinical trials, BLISS-52 and BLISS-76.
3. Objective three is a single centre prospective study.

Study Population and Sampling Methods:

Objective I patient selection: Patients with active disease, SLEDAI-2K ≥0, will be identified in the TLC database. All patients must have follow up visits at 3 and 6 months.

Objective II: Data from BLISS-52 and BLISS-76 trials will be used. Objective III patient selection: Patients followed at the Toronto Lupus Clinic from May 2017 to December 2017. Patients will be identified based on active disease with a flare (increase in SLEDAI-2K by at least 4 requiring an increase in the dose of prednisone to ≥ 15 mg/day or initiation of prednisone at ≥ 15 mg/day).

Objective III patient selection: Patients followed at the Toronto Lupus Clinic from May 2017 to December 2017. The investigator will identify patients with active disease with a flare (increase in SLEDAI-2K by at least 4 requiring an increase in the dose of prednisone to ≥ 15 mg/day or initiation of prednisone at ≥ 15 mg/day).

Data Sources:

The University of Toronto Lupus Cohort dataset and GSK BLISS-52 and BLISS-76 trial data The Toronto Lupus Cohort (TLC) is the largest lupus cohort in Canada, and more than 1600 patients have been enrolled in this cohort. Patients in the TLC are seen at regular intervals (2-6 months apart) and data, including laboratory and clinical parameters important to lupus, is collected using a well-defined protocol.

Data Analysis Methods:

In objective I - Phase 1 will focus on the identification of scenarios of real patients to derive weight scores for Glucocorticosteroid (GCS). Phase 2 will focus on the development of SLEDAI-2KG (derivation of an equation to explain the link between SLEDAI-2K and GCS doses) and phase 3 focused on SLEDAI-2KG validation.

The analysis of the initial validation of SLEDAI-2KG will be conducted on the selected patients from the TLC. Improved patients (responders) will be identified based on SLEDAI-2K definition of improvement and further will be studied by calculating the SLEDAI-2KG using the above described models. The mean change of SLEDAI-2K scores and the mean change of SLEDAI-2KG scores in the responders will be studied. Using the SLEDAI-2K responders as "Gold Standard", it will be determined if SLEDAI-2KG responders are true responders and not false responders.

Concurrent construct validity: A clinician (external construct) who does not know the patients and will evaluate each patient's record (electronic record and medical chart) and assign a clinical activity score for each assessment according to the following scale: improved, same, and worse, using standardized predefined definitions. The correlation between the external construct and the change in SLEDAI-2K and SLEDAI-2KG scores will be studied. Using the clinician scoring of disease activity-Improved as "Gold Standard", the results of SLEDAI-2K and SLEDAI-2KG responders will be analyzed by constructing two 2x2 tables.

Sample Size for 3 objectives:

Sample Size 1: The sample size calculation of needed scenarios was based on the assumption of reliability (Intra-class Correlation Coefficient (ICC)) ≥ 0.80 with a standard error of 0.05 and 3 raters. The required minimum was 46 scenarios.

Sample Size 2: For objective two all data available from the BLISS-52 and BLISS-76 trials will be used.

Sample Size 3: For objective three the investigator's target sample size is 100 patients and to achieve this number at least 18 months will be required and subsequently a 6 months period for follow-up for each patients. Based on the COSMIN recommendations, a sample size ≥100 is recommended in this step

ELIGIBILITY:
Inclusion Criteria:

Objective I:

* ≥4 American College of Rheumatology (ACR) criteria or 3 ACR criteria plus a typical histological lesion of SLE on renal or skin biopsy
* Clinician's diagnosis based on his/her assessment
* Patients from the Toronto Lupus Clinic with regular follow-up, defined as having follow up visits at 3 and 6 months from the baseline visit (1st study visit).

Objective II:

• Participant in the BLISS-52 and BLISS-76 trials

Objective III:

* ≥4 American College of Rheumatology (ACR) criteria or 3 ACR criteria plus a typical histological lesion of SLE on renal or skin biopsy
* Increase in SLEDAI-2K ≥4
* Clinician's diagnosis based on his/her assessment

Exclusion Criteria:

Objective I and III:

* Patients with missing follow up visits at 3 and 6 months from the baseline visit (1st study visit).
* Patients with missing data in the charts for all visits.

Objective II:

• Participants who did not complete the trial and therefore have missing data points for primary endpoint measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Objective I Initial Development and Validation of SLEDAI-2KG This is a retrospective validation study of SLEDAI-2KG using the University of Toronto Lupus Clinic (TLC) database. Clinical and laboratory data is collected according to a standard protocol at regular intervals (2 to 6 months between visits) and stored on a computer database.
  Objective II Further retrospective validation of SLEDAI-2KG using BLISS trial data.
  All patients in GSK BLISS-52 (N=865) and BLISS-76 (N=819) were assessed at regular intervals and data including clinical and laboratory features of SLE, medications and in particular corticosteroids was collected and will be used in the validation of SLEDAI-2KG.
  Objective III Assessment of concurrent construct validity of SLEDAI-2KG prospectively in the TLC Cohort Patients from the TLC with active disease with a flare (increase in SLEDAI-2K by at least 4) that requires an increase in the dose of prednisone to ≥15 mg/day or initiation of prednisone at ≥15 mg/day.
Sampling Method: Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Objective I - Initial Development and Validation of Systemic Lupus Erythematosus Disease Activity Index-2000 Glucocorticosteroid (SLEDAI-2KG) | 3 months
  The new index SLEDAI-2KG will be validated against the old index Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) in the TLC cohort. Improved patients (responders) will be identified based on SLEDAI-2K definition of improvement (decrease in the total score by ≥4).
  Clinician scoring on a Likert scale (external construct) for disease activity - Improvement based on predefined definitions
Objective II - Further validation of Systemic Lupus Erythematosus Disease Activity Index-2000 Glucocorticosteroid (SLEDAI-2KG) using BLISS trial data | 5 months
  SLEDAI-2KG will be further validated using BLISS-52 and BLISS-7S trial data on all patients that were enrolled. The primary endpoint in both trials was SLE Responder Index (SRI). The SRI incorporates the Safety of Estrogens in Lupus Erythematosus-National Assessment-SLEDAI (SELENA-SLEDAI), British Isles Lupus Assessment Group (BILAG), and Physician Global Assessment (PGA). The primary outcome of this objective is the SRI-modified: The SRI-modified will include the 2nd and 3rd components of SRI, but replace the SELENA-SLEDAI with the SLEDAI-2KG.
Objective IIIA - Assessment of concurrent construct validity of Systemic Lupus Erythematosus Disease Activity Index-2000 Glucocorticosteroid (SLEDAI-2KG) prospectively in the University of Toronto Lupus Clinic | 8 months
  Improved patients (responders) will be identified based on Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) definition of improvement (decrease in the total score by ≥4).
Objective IIIB - Identification of Systemic Lupus Erythematosus Disease Activity Index-2000 Glucocorticosteroid (SLEDAI-2KG) Responders | 8 months
  SLEDAI-2KG improved patients (responders) will be identified based on the definition of improvement (decrease in the total score by ≥4).

CONTACTS AND LOCATIONS:
Overall Officials: Zahi Touma, MD PhD, Principal Investigator — University Health Network and University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No